CLINICAL TRIAL: NCT03062787
Title: Early Effect of Cingal® Compared to Monovisc® in Patients With Osteoarthritis of the Knee (EEFFEK Study)
Brief Title: Early Effect of Cingal® Compared to Monovisc® in Patients With Osteoarthritis of the Knee
Acronym: EEFFEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmascience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN-401
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cingal® (Experimental): Single 4 ml intra-articular injection of Hyaluronic Acid plus Triamcinolone Hexacetonide
  Interventions: Device: Cingal® (Hyaluronic Acid plus Triamcinolone Hexacetonide)
- Monovisc® (Active Comparator): Single 4 ml intra-articular injection of Sodium Hyaluronate
  Interventions: Device: Monovisc® (Sodium hyaluronate)

INTERVENTIONS:
Device: Cingal® (Hyaluronic Acid plus Triamcinolone Hexacetonide) — Intra-articular injection
  Other Names: Cingal®
  Arms: Cingal®
Device: Monovisc® (Sodium hyaluronate) — Intra-articular injection
  Other Names: Monovisc®
  Arms: Monovisc®

SUMMARY:
It is a post-license, multicenter, randomized, single blind, controlled study comparing a single injection of Cingal® (study arm) with a single injection of Monovisc® (control arm).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Diagnosed with osteoarthritis of the knee
* Candidate for an intra-articular injection (single joint, unilateral) of Monovisc® or Cingal® as part of their routine clinical care and in accordance with the locally approved label

Exclusion Criteria:

* Previous intra-articular injection within the last 6 months from enrolment
* Known hypersensitivity to cortico-steroids, hyaluronic acid or any component of Cingal® or Monovisc®
* Infectious, traumatic or neoplasic component of knee pathology
* Surgery of the knee within the last 6 months or scheduled surgery in the next two months from enrolment
* Patients with impaired cardio-renal function, endocrine, or other diseases or conditions that use of corticosteroid is warned.
* Patients with known bleeding disorders
* Patient currently treated with oral steroids or opioids
* Patients that, in the investigators' opinion, are unlikely to comply with protocol
* Pregnant or nursing women or women who suspect they might be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Compare the local pain reduction after a single injection of Cingal® or Monovisc® over a 6 weeks period in patients with osteoarthritis of the knee assessed with the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 6 weeks post injection
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)

SECONDARY OUTCOMES:
Compare the maximum pain reduction by treatment arm | 6 weeks post injection
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Compare the time to maximum pain reduction by treatment arm | 6 weeks post injection
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Change in stiffness and physical function | 6 weeks post injection
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Overall change of WOMAC score | 6 weeks post injection
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Time to maximum WOMAC score reduction | 6 weeks post injection
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, PhD, Principal Investigator — McMaster University
Locations (5):
- Canada (5):
  - Site 04, Barrie, Ontario
  - Site 03, Hamilton, Ontario
  - Site 02, Kanata, Ontario
  - Site 05, Laval, Quebec
  - Site 01, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No